CLINICAL TRIAL: NCT01615653
Title: Prospective Randomized Trial of EUS Guided Celiac Ganglia Neurolysis (CGN) Versus EUS Guided Celiac Plexus Neurolysis (CPN) for Pancreatic Cancer Pain
Brief Title: EUS Guided Celiac Neurolysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: American College of Gastroenterology (Other)
Responsible Party: Principal Investigator, Michael Levy, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09-005037
Record Dates: First submitted 2012-04-17; First posted 2012-06-08 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Pancreatic Cancer Pain
Keywords: Pancreatic cancer; Pancreas cancer; Pain; Celiac Plexus; Neurolysis
MeSH Terms: conditions — Pancreatic Neoplasms; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EUS 1 (Active Comparator)
  Interventions: Procedure: EUS
- EUS 2 (Active Comparator)
  Interventions: Procedure: EUS

INTERVENTIONS:
Procedure: EUS — EUS Guided Therapy

SUMMARY:
* Hypothesis:

  - Direct CGN enhances neurolytic drug delivery into celiac ganglia and increases the efficacy of neurolysis and subsequent pain control and survival in patients with pancreatic carcinoma.
* Rationale:

  * Standard CPN leads to inaccurate delivery of the injectate with rapid dispersal thereby only briefly remaining in contact with neural structures and limiting the degree of neurolysis. Poor targeting and delivery of a neurolytic agent may result in diminished neurolysis and decrease efficacy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Unresectable pancreatic carcinoma (T4 or M1) or advanced T3 disease
* 2. Cytologic or histologic confirmation of pancreatic carcinoma
* 3. Abdominal pain (≥ 3 on NRS scale), ≥ 2 days/week, lasting ≥ 1 hour/ day, stable intensity for ≥ 7 days
* 4. EUS clinically indicated (for non-study purposes)

Exclusion Criteria:

* 1. Uncorrectable coagulopathy: (INR) > 1.5 and/or platelets < 50,000
* 2. Abdominal surgery within 1 month
* 3. Prior celiac plexus or ganglia neurolysis.
* 4. Initiation or modification in chemotherapy or radiotherapy within prior 7 days.
* 5. Direct tumor infiltration of the celiac trunk and/or celiac ganglia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Pain assessed using a numerical rating scale (NRS) from 0 to 10. | Baseline to 6 months
  pain response will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Levy MJ, Gleeson FC, Topazian MD, Fujii-Lau LL, Enders FT, Larson JJ, Mara K, Abu Dayyeh BK, Alberts SR, Hallemeier CL, Iyer PG, Kendrick ML, Mauck WD, Pearson RK, Petersen BT, Rajan E, Takahashi N, Vege SS, Wang KK, Chari ST. Combined Celiac Ganglia and Plexus Neurolysis Shortens Survival, Without Benefit, vs Plexus Neurolysis Alone. Clin Gastroenterol Hepatol. 2019 Mar;17(4):728-738.e9. doi: 10.1016/j.cgh.2018.08.040. Epub 2018 Sep 12. PMID 30217513